CLINICAL TRIAL: NCT03331211
Title: Observation of the Effect of Chemotherapy Combined With Tyrosinase Inhibitor on the Reactivation of CMV and EBV in Patients With Acute Lymphoblastic Leukemia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Principal Investigator, Qifa Liu, Professor, Nanfang Hospital, Southern Medical University
Other Study IDs: NFH-ALL-CMV-2017
Record Dates: First submitted 2017-10-31; First posted 2017-11-06 (Actual); Last update posted 2017-11-08 (Actual); Status verified 2017-09

CONDITIONS: Leukemia, Lymphoblastic, Acute
Keywords: Leukemia, Lymphoblastic, Acute
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Dasatinib; nilotinib; ponatinib; Imatinib Mesylate

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Chmotherapy combined with TKIs: Patients with ALL were treated by chmotherapy and TKIs(PDT-NFH-2016)
  Interventions: Drug: TKIs

INTERVENTIONS:
Drug: TKIs — Dasatinib combined with Chematherapy
  Other Names: Dasatinib; Nilotinib; Ponatinib; Imatinib

SUMMARY:
Philadelphia-chromosome-positive or partial ph-like acute lymphoblastic leukemia (ALL) preferred chemotherapy combined with tyrosine kinase inhibitors (TKIS) therapy. Recently we found that there were cytomegalovirus reactivation and even cytomegalovirus infection in three ALL patients treated with chemotherapy combined with TKIs. However, the cytomegalovirus risk after dasatinib use in patients with philadelphia-chromosome-positive ALL is still unknown. It is reported that dasatinib can be observed in the treatment of philadelphia-chromosome-positive leukemia patients with significant increase in large granular lymphocytes, the cytomegalovirus is often positive, and this part of the patient's prognosis is relatively good. Dasatinib can inhibit SRC and TEC kinase, and induce immune function inhibition,and in vitro experiments have confirmed that it inhibits the immune function of T cells and NK cells. In this study, we examined the potential association between cytomegalovirus AND EBV reactivation the treatment of chemotherapy combined with TKIs, and the numbers of large granular cells and NK cell activity.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with acute lymphoblastic leukemia who had not previously received chemotherapy (except for hormone preconditioning) or started with chemotherapy but not more than 3 days, and CMV and EBV quantitative negative;
2. Age Limits:>or= 14 years old.

Exclusion Criteria:

1. Patients who had previously received chemotherapy and hematopoietic stem cell transplantation;
2. Patients with CMV and EBV infection before treatment and not to turn yin;
3. The researchers considered unsuitable patients.

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnosed with acute lymphoblastic leukemia who had not previously received chemotherapy (except for hormone preconditioning) or started with chemotherapy but not more than 3 days, and CMV and EBV quantitative negative.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2017-11-01 (Actual); Primary Completion 2019-09-01 (Estimated); Study Completion 2019-09-01 (Estimated)

PRIMARY OUTCOMES:
CMV and EBV reactivation rate | 2 years
  Evaluation of CMV and EBV reactivation after chemotherapy combined with TKIs therapy in ALL patients

SECONDARY OUTCOMES:
The number of large granulosa cells and T、B、NK cell activity | 2 years
  Evaluation of the relationship between the number of large granulosa cells and T、B、NK cell activity in patients with CMV positive after TKIs therapy

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Hematology,Nanfang Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ishiyama K, Kitawaki T, Sugimoto N, Sozu T, Anzai N, Okada M, Nohgawa M, Hatanaka K, Arima N, Ishikawa T, Tabata S, Onaka T, Oka S, Nakabo Y, Amakawa R, Matsui M, Moriguchi T, Takaori-Kondo A, Kadowaki N. Principal component analysis uncovers cytomegalovirus-associated NK cell activation in Ph+ leukemia patients treated with dasatinib. Leukemia. 2017 Jan;31(1):203-212. doi: 10.1038/leu.2016.174. Epub 2016 Jun 14. PMID 27349810